CLINICAL TRIAL: NCT05519371
Title: Efficacy and Safety Evaluation of Injectable Remimazolam for Intraoperative Arousal in Scoliosis Orthopedics
Brief Title: Remimazolam and Scoliosis Orthopedics
Acronym: rimazolam
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Anshi Wu, Director of department of anesthesiology, Chaoyang Hospital, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20220817
Record Dates: First submitted 2022-08-16; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Benzodiazepines
MeSH Terms: interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remimazolam group (Experimental): For induction of anesthesia, rimazolam benzoate was pumped at a rate of 12 mg/kg/h; for maintenance of anesthesia, 1.0-2.0 mg/kg/h rimazolam was given as a continuous pump.
  Interventions: Drug: Remimazolam
- propoful group (Active Comparator): For induction of anesthesia, propofol medium-length chain fatty milk injection 2 mg/kg was given by intravenous push; for maintenance of anesthesia, 6-8 mg/kg/h propofol medium-length chain fatty milk injection was given by continuous pumping.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — During induction of anesthesia, the rimazolam group was given rimazolam pumped at a rate of 12 mg/kg/h
  During the maintenance phase of anesthesia, the rimazolam group was given 1.0-2.0 mg/kg/h of rimazolam continuously pumped.
  Arms: remimazolam group
Drug: Propofol — During induction of anesthesia, propofol 2mg/kg was given, and during the maintenance phase of anesthesia, propofol 6-8mg/kg/h was given as a continuous pump.
  Arms: propoful group

SUMMARY:
Spinal cord injury is one of the most dangerous complications of scoliosis orthopedic surgery, and the Stagnara awakening test has been used in orthopedic spine surgery and is considered the "gold standard" for detecting spinal cord injury. During the awakening test, the patient is awakened from anesthesia and, in conjunction with a neurological assessment, moves his or her fingers and toes to determine the integrity of spinal cord motor function in order to avoid spinal cord injury. During this procedure, the patient still requires a degree of sedation and analgesia to tolerate tracheal intubation and surgical pain. Remazolam benzoate for injection is a new class of benzodiazepines that are ultra-short-acting sedative/anesthetic drugs. It has the advantages of rapid onset, rapid elimination, and no drug accumulation by continuous infusion, and has the advantage of being applied to wake up during spinal orthopedic surgery, but its effectiveness and safety are still unclear. This study aims to elucidate the safety and efficacy of rimazolam benzoate for injection for arousal in spinal orthopedic surgery through a single-center, randomized, single-blind, positive drug-controlled trial, with the aim of providing a basis for the development of a safe and effective anesthetic protocol for such surgery.

ELIGIBILITY:
Criteria:

Inclusion Criteria:

1. Age greater than 18 years and less than 60 years
2. Elective scoliosis orthopaedic surgery under general anesthesia.
3. ASA Physical Score I-III
4. Signed informed consent.

Exclusion Criteria:

1. Patients who cannot understand the method and requirements of the arousal test and cannot cooperate in completing the arousal test.
2. Patients with limb sensory-motor dysfunction.
3. Patients with a history of severe neurological disorders.
4. Patients with psychiatric disorders.
5. Patients who have taken benzodiazepines and/or opioids daily for one month or intermittently for the last three months.
6. Patients with concomitant severe respiratory and circulatory disorders, including acute heart failure, unstable angina, resting ECG heart rate <50 beats/min, QTc: ≥ 470ms in men and ≥ 480ms in women, third-degree AV block, severe arrhythmia, moderate to severe heart valve disease, chronic obstructive pulmonary disease, and history of asthma.
7. Abnormal liver and kidney function: ALT and/or AST exceeding 2.5 times the upper limit of the medical reference range; urea or urea nitrogen ≥1.5 × ULN, blood creatinine greater than the upper limit of normal values.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Mean time to arousal | Perioperative period
  the time between the cessation of intraoperative drug infusion and the subject's ability to move the toes on command.

SECONDARY OUTCOMES:
Quality of arousal | Perioperative period
  Class I: the patient wakes up when called, is quiet and moves the limbs as instructed; Class II, the patient wakes up suddenly, moves the limbs involuntarily, does not endanger the internal fixation and tracheal tube, and can move the limbs as instructed; Class III, the patient wakes up suddenly, moves the trunk violently and requires pressure to not endanger the internal fixation and tracheal tube
Proportion of successful induction of anesthesia | Perioperative period
  The criteria for successful induction of anesthesia were that both of the following two requirements were met: completion of tracheal intubation; and no use of remedial sedative drugs
Mean time from initiation of dosing to MOAA/S score ≤1 | Perioperative period
  Mean time from initiation of dosing to MOAA/S score ≤1
Mean time from discontinuation at the end of surgery to full awakening of the subject | Perioperative period
  time to the first of three consecutive MOAA/S scores of 5
EEG characteristics during the induction, maintenance and awakening periods | Perioperative period
  EEG power in alpha band, beta band, theta band, and gamma band

OTHER OUTCOMES:
Other adverse events | Postoperative 28 days
  Other adverse events within 28 days after surgery were noted

IPD SHARING:
Plan to Share IPD: No